CLINICAL TRIAL: NCT01851265
Title: A Two-part, Randomised, Open-label, Multicentre, Phase I Study to Determine the Effect of Food on the Pharmacokinetics of Olaparib Following Single 400 mg Doses of the Capsule Formulation in Patients With Advanced Solid Tumours.
Brief Title: D081AC00001 Food Interaction With Olaparib Capsule in Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: D081AC00001; 2013-001255-13 (EudraCT Number)
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Solid Tumours
Keywords: oncology, cancer, tumour, neoplasm, anticancer drug, food effect, area under the curve, pharmacokinetics, olaparib, solid tumour, metabolites, drug availability
MeSH Terms: conditions — Neoplasms | interventions — olaparib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fasted (Other): Olaparib capsules following no breakfast
  Interventions: Drug: Olaparib; Other: Dietary Fasted
- Standard meal (Other): Olaparib capsules after standard breakfast
  Interventions: Drug: Olaparib; Other: Dietary standard
- High Fat (Other): Olaparib capsules after high fat breakfast
  Interventions: Drug: Olaparib; Other: Dietary High Fat

INTERVENTIONS:
Drug: Olaparib — 400mg olaparib capsule formulation taken 30 minutes after allocated meal. 5-14 days between arms.
Other: Dietary Fasted — Allocated breakfast prior to dosing with 400mg olaparib capsules
  Arms: Fasted
Other: Dietary standard — Allocated breakfast prior to dosing with 400mg olaparib capsules
  Arms: Standard meal
Other: Dietary High Fat — Allocated breakfast prior to dosing with 400mg olaparib capsules
  Arms: High Fat

SUMMARY:
This is a 2 part study for patients with solid tumours. The purpose of Part A is to measure the amount of olaparib or its breakdown products in the bloodstream for up to 72 hours after eating 3 different breakfasts (high calorie, regular and none). In Part B Patients can take olaparib capsules daily and study assessments will be recorded for 6 months (minimum). Treatment can continue for as long as the patient is benefitting. Throughout the study patients will be monitored for any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years, male and female
* Able to eat a high-fat breakfast within a 30-minute period, as provided by the study site
* Histologically or, where appropriate, cytologically confirmed malignant solid tumour refractory or resistant to standard therapy and for which no suitable effective standard therapy exists
* ECOG performance status ≤2
* Normal organ and bone marrow function measured within 28 days prior to administration of IP as defined in protocol

Exclusion Criteria:

* Participation in another clinical study with an IP during the last 14 days (or a longer period depending on the defined characteristics of the agents used)
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 2 weeks prior to study treatment (or a longer period depending on the defined characteristics of the agents used).
* Toxicities (≥CTCAE Grade 2) caused by previous cancer therapy, excluding alopecia
* Patients unable to fast for up to 14 hours or who have type I or type II diabetes
* Patients who have gastric, gastro-oesophageal or oesophageal cancer

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-07-04 (Actual); Primary Completion 2013-10-18 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Olaparib (Cmax and tmax) | Blood samples will be collected in each of the 3 treatment periods in Part A at these time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72hours post dose
  Rate and extent of absorption of olaparib following single-dose olaparib by assessment of maximum plasma olaparib concentration (Cmax) and time to reach maximum plasma concentration (tmax)
Pharmacokinetics of Olaparib (AUC0-t) | Blood samples will be collected in each of the 3 treatment periods in Part A at these time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72hours post dose.
  Rate and extent of absorption of olaparib following single-dose olaparib by assessment of area under the plasma concentration time curve from zero to the last measurable time point (AUC0-t)
Pharmacokinetics of Olaparib (AUC) | Blood samples will be collected in each of the 3 treatment periods in Part A at these time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72hours post dose
  Rate and extent of absorption of olaparib following single-dose olaparib by assessment of area under the plasma concentration time curve from zero to infinity (AUC)
Pharmacokinetics of Olaparib Pharmacokinetics of Olaparib (CL/F, Vz/F, λz and t½) | Blood samples will be collected in each of the 3 treatment periods in Part A at these time points: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72hours post dose.
  Rate and extent of absorption of olaparib following single-dose olaparib by assessment of apparent clearance following oral administration (CL/F), apparent volume of distribution (Vz/F), terminal rate constant (λz), and terminal half-life (t½)

SECONDARY OUTCOMES:
Safety monitoring of Olaparib | AEs will be collected from signed informed consent up to 30-day post last dose in Part A. For patients in Part B, AE's will be collected until the final patient has completed 6 months in Part B, including 30 day follow up for those who discontinue
  Assessment of adverse events (AEs), graded by CTCAE (v4.0), physical examination, vital signs (including BP and pulse), standard 12-lead ECG and evaluation of laboratory parameters (clinical chemistry, haematology, and urinalysis). Assessment of physical examination, vital signs, ECG and evaluation of laboratory parameters will occur at screening, on the day before dosing in each treatment period and 30 days after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Anitra Fielding, Study Director — AstraZeneca Senior Research Physician; Christian Rolfo, Principal Investigator — UZ Antwerpen; Wendy Bannister, Study Chair — AstraZeneca Study Statistician
Locations (7):
- Belgium (3):
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Wilrijk
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht
- United Kingdom (2):
  - Research Site, Glasgow
  - Research Site, Manchester

REFERENCES:
- See also: D081AC00001_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1820&filename=D081AC00001_Study_Synopsis.pdf